CLINICAL TRIAL: NCT05699993
Title: An Open-label, 2-cycle Clinical Study to Evaluate the Drug Interaction Between Itraconazole or Dextromethorphan and IBI351 in Healthy Subjects
Brief Title: A Study of IBI351 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIBI351P003
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Itraconazole; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI351+ itraconazole (Other): Enrolled subjects were treated with IBI351 on an empty stomach on Day 1. Itraconazole was administered orally once daily after a standardized meal from Day 3 to Day 6. IBI351 and itraconazole were administered simultaneously on an empty stomach on Day 7. On Day 8, itraconazole was orally administered once after a standard meal.
  Interventions: Drug: Itraconazole; Drug: IBI351
- IBI351+ dextromethorphan (Other): Enrolled subjects were orally administered dextromethorphan on an empty stomach on Day 1. IBI351 and dextromethorphan were orally administered simultaneously on an empty stomach on Day 3, followed by IBI351 12 hours later.
  Interventions: Drug: IBI351; Drug: Dextromethorphan

INTERVENTIONS:
Drug: Itraconazole — Itraconazole was administered orally
  Arms: IBI351+ itraconazole
Drug: IBI351 — IBI351 was administered orally
Drug: Dextromethorphan — Dextromethorphan was administered orally
  Arms: IBI351+ dextromethorphan

SUMMARY:
This is an open-label, two-cycle clinical study to evaluate the drug interaction between itraconazole or dextromethorphan and IBI351 in healthy subjects. A total of two cohorts of 12 healthy male subjects were planned to be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the trial, fully understand the content, process and possible adverse reactions of the trial, and be able to complete the study according to the requirements of the trial protocol.
2. Healthy male subjects aged 18 to 45 years (including both ends) at the time of signing informed consent.
3. Body weight is not less than 50 kg, and body mass index (BMI) is in the range of 19 ~ 26 kg/m2 (including both ends).
4. Physical examination, vital signs, routine laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function), thyroid function, 12-lead electrocardiogram, chest CT, abdominal ultrasound (hepatobiliary, pancreatic, spleen and kidney), echocardiography (only applicable to Cohort 1 subjects) showed no abnormalities; or abnormal test results but judged as normal or clinically insignificant by the investigator.

Exclusion Criteria:

1. have taken any products containing alcohol or have a positive alcohol breath test (≥ 20 mg/100 ml) within 24 hours before taking study medication.
2. hepatitis B surface antigen HBsAg positive.
3. hepatitis C virus antibody positive.
4. positive AIDS antigen/antibody or Treponema pallidum antibody.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
maximum concentrations (Cmax ) for IBI351 | approximately 10 days
maximum concentrations (Cmax ) for dextromethorphan | approximately 10 days
area under the curve from time 0 to infinity(AUC0-inf) for IBI351 | approximately 10 days
area under the curve from time 0 to infinity(AUC0-inf) for dextromethorphan | approximately 10 days

SECONDARY OUTCOMES:
time-to-maximum concentration (Tmax) for IBI351 | approximately 10 days
half-life (t1/2) for IBI351 | approximately 10 days
area under the curve from time 0 to time (AUC0-t) for IBI351 | approximately 10 days
apparent clearance (CL/F) for IBI351 | approximately 10 days
apparent volume of distribution(Vz/F) for IBI351 | approximately 10 days
time-to-maximum concentration (Tmax) for dextromethorphan | approximately 10 days
half-life (t1/2) for dextromethorphan | approximately 10 days
area under the curve from time 0 to time (AUC0-t) for dextromethorphan | approximately 10 days
apparent clearance (CL/F) for dextromethorphan | approximately 10 days
apparent volume of distribution(Vz/F) for dextromethorphan | approximately 10 days
area under the curve for dextrorphan | approximately 10 days
maximum concentrations (Cmax ) for dextrorphan | approximately 10 days
number of participants with abnormal hematology tests | approximately 10 days
number of participants with abnormal chemistry parameters | approximately 10 days
number of participants with abnormal vital signs | approximately 10 days
number of participants with abnormal physical examination findings | approximately 10 days
number of participants with abnormal ECG readings | approximately 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China